CLINICAL TRIAL: NCT04778579
Title: Phase 2 Study of the Infusion of Differentiated Autologous T-cells From Peripheral Blood, Expanded and Transduced With a Lentivirus to Express a Chimeric Antigen Receptor With Anti-CD19 Specificity (A3B1) Conjugated With the Co-stimulatory Regions 4-1BB and CD3z (ARI-0001 Cells) in Patients With CD19+ Acute Lymphoid Leukemia Resistant or Refractory to Therapy
Brief Title: Study of the Infusion of ARI-0001 Cells in Patients With CD19 + Acute Lymphoid Leukemia Resistant or Refractory to Therapy
Acronym: CART19-BE-02
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sara V. Latorre (Other)
Collaborators: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Sara V. Latorre, Clinical Research Manager, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Organization: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART19-BE-02
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Acute Lymphoid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — CTL019 chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARI-0001 (Experimental): After pretreatment, adult differentiated autologous T-cells with a chimeric antigen receptor with anti-CD19 specificity will be transfused.
  Interventions: Drug: ARI-0001 cells

INTERVENTIONS:
Drug: ARI-0001 cells — Adult differentiated autologous T-cells from peripheral blood, expanded and transduced with a lentivirus to express a chimeric antigen receptor with anti-CD19 specificity (A3B1) conjugated with the co-stimulatory regions 4-1BB and CD3z
  Other Names: CART19; PEI 19-187

SUMMARY:
To assess the efficacy (in terms of response rate and duration) of the infusion of ARI-0001 cells (Adult differentiated autologous T-cells from peripheral blood, expanded and transducted with a lentivirus to express a chimeric antigen receptor with anti-CD19 specificity [A3B1] conjugated to the 4-aBB and CD3z co-stimulatory regions) in patients with resistant or refractory CD19+ acute lymphoid leukemia

ELIGIBILITY:
Inclusion Criteria:

1. Diagnoses of CD19+ acute lymphoid leukemia, with a life expectancy of less than 2 years that meet the following conditions:

   1. Relapsed/refractory not candidate for transplantation (due to associated diseases or absence of donor)
   2. in allogenic post-transplant relapse.
2. Measurable disease understood as the presence of measurable residual disease by flow cytometry in bone marrow or peripheral blood
3. Age less than 70 years (from 18 to 70).
4. ECOG functional status from 0 to 2
5. Life expectancy of at least 3 months.
6. Adequate venous access to perform a lymphapheresis. Absence of contraindications for it.
7. Signature of informed consent.

Exclusion Criteria:

1. Treatment with any experimental or non-marketed substance within four weeks prior to recruitment, or actively participating in another therapeutic trial.
2. Previous treatment with CART therapy (commercial or experimental)
3. Diagnosis of another neoplasm, past or present. Patients may be included in complete remission for more than 3 years, or have a history of non-melanoma skin cancer or in-situ carcinoma resected completely.
4. Relief of central nervous system (CNS-3) at the time of inclusion. Inclusion will be permitted in patients with a lower grade (CNS-2) or CNS-3 who have responded to intrathecal chemotherapy.
5. Isolated extramedullary involvement (i.e. in the absence of minimal residual disease in peripheral blood, bone marrow, or cerebrospinal fluid)
6. Early relapse after transplantation (less than 3 months for mononuclear cell apheresis, less than 6 months for infusion of ARI-0001)
7. Active immunosuppressive treatment for graft-versus-host disease and other diseases. The use of corticosteroids to control leukaemia at the time of inclusion should be limited as much as possible and should be discontinued prior to infusion of ARI-0001 cells.
8. Active infection requiring systemic medical treatment such as chronic kidney infection, chronic lung infection or tuberculosis.
9. HIV infection.
10. Positive serology for hepatitis B, defined as a positive test for HBsAg. In addition, if the patient is HBsAg negative but has anti-HBc antibodies it will be necessary to perform a DNA test of the hepatitis B virus, and if the result is positive the patient will be excluded
11. Positive serology for hepatitis C, defined as a positive test for anti-VHC antibodies confirmed by RIBA
12. Concurrent uncontrolled medical illnesses including cardiac, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological or psychiatric diseases that in the opinion of the investigator are potential risk factors to the patient.
13. Severe organ involvement, defined as cardiac ejection fraction <40%; DLCO <40%; calculated glomerular filtrate <30 ml/min; or bilirubin > 3 times the upper limit of normality (unless Gilbert syndrome).
14. Pregnant or lactating women. Woman of childbearing potential should have a negative pregnancy test in the screening phase.
15. Women of childbearing potential, including those whose last menstrual cycle was in the year prior to screening, who are unable or unwilling to use highly effective contraceptive methods* from the start of the study to the completion of the study.
16. Men who cannot or do not wish to use highly effective contraceptive methods* from the beginning of the study until the end of the study

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | 20 days after infusion
  • Response rate with measurable residual disease negative by multiparametric flow cytometry

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico Universitario Virgen de La Arrixaca, Murcia
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital U. Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ortiz-Maldonado V, Martinez-Cibrian N, Alserawan L, Espanol-Rego M, Navarro-Velazquez S, Albiol N, Oliver-Caldes A, Triguero A, Herrero-Garcia M, Gutierrez-Herrero S, Benitez-Ribas D, Paciello ML, Torrent A, Delgado-Serrano J, Sanchez-Castanon M, Calderon H, Mata JJ, Sanchez-Salinas A, Saez-Penataro J, Sans-Pola C, Calvo-Orteu M, Lopez-Corral L, Kwon M, Rifon J, Charry P, Alonso-Fernandez RA, Huguet M, Blazquez-Goni C, Sanchez-Pina JM, Sanchez R, Rosa-Rosa JM, Martinez-Lopez J, Blanquer M, Ribera JM, Urbano-Ispizua A, Bachiller M, Palau L, Olesti E, Calvo G, Martin-Martin L, Orfao A, Gonzalez-Navarro EA, Domenech G, Varea S, Juan M, Delgado J, Esteve J. Varnimcabtagene autoleucel for adults with relapsed or refractory B-cell precursor acute lymphoblastic leukaemia in Spain (CART19-BE-02): a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2026 Feb 3:S2352-3026(25)00328-X. doi: 10.1016/S2352-3026(25)00328-X. Online ahead of print. PMID 41651004